CLINICAL TRIAL: NCT05482737
Title: Clinical Impact of Red Cell Storage Age: Individual Patient Data Meta-Analysis of Four Recent Large Randomized Trials
Brief Title: Clinical Impact of Red Cell Storage Age
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: Pending 4
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: RBC Transfusions
Keywords: RBC transfusions; storage age; meta-analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Reference group: Transfused RBC stored 8-35 days
  Interventions: Other: no intervention
- less than or equal 7 days: Transfused RBC stored =<7 days
  Interventions: Other: no intervention
- more than 7 days: Transfused RBC stored <7 days
  Interventions: Other: no intervention
- less that or equal 10 days: Transfused RBC stored =<10 days
  Interventions: Other: no intervention
- more that 10 days: Transfused RBC stored >10 days
  Interventions: Other: no intervention
- more than 35 days: Transfused RBC stored >35 days
  Interventions: Other: no intervention
- less than or equal 35 days: Transfused RBC stored =<35 days
  Interventions: Other: no intervention
- less than 18 days: Transfused RBC stored <18 days
  Interventions: Other: no intervention
- more than or equal 18 days: Transfused RBC stored =>18 days
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is an observational retrospective study (meta-analysis)

SUMMARY:
The recent four RCTs evaluating effects of RBC storage age on morbidity and mortality found no statistically significant adverse effects of longer stored RBC compared to shorter storage ages. Unfortunately, none of these RCTs had sufficient numbers of subjects receiving RBC at either storage age extreme to identify consequences of RBC transfusion at these limits. To better investigate effects of RBC storage age on clinical outcomes, this study will perform secondary meta-analyses of merged common patient data elements -individual patient data (IPD) meta-analysis (IPDMA) - from the nearly 33,000 subjects enrolled in the four RCTs.

ELIGIBILITY:
Inclusion Criteria:

* Received at least one RBC transfusion
* >=18 years of age

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects in the recent four RCTs who are 18 years or older and have received at least one RBC transfusion.
Sampling Method: Non-Probability Sample
Enrollment: 33000 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 28 days after transfusion
  Estimate the effect of transfused RBC storage-age on time to all-cause mortality
Hospital length of stay | after transfusion through 28 days
  Estimate the effect of transfused RBC storage-age on hospital stay

SECONDARY OUTCOMES:
All-cause mortality at 28 days for long-storage | 28 days after transfusion
  all-cause mortality at 28 days comparing subjects who received (one or more) RBC unit ≥ 35 days vs. no unit > 35 days
28 day mortality for short-storage | 28 days after transfusion
  28 day mortality for subjects who received (one or more) RBC unit ≤ 7 days vs. no unit ≤ 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Marie Steiner, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided